CLINICAL TRIAL: NCT00848263
Title: Unstable Fractures of the Distal Radius: Randomised Controlled Trial of Volar Plate Versus Dorsal Nail Plate Fixation.
Brief Title: Unstable Fractures of the Distal Radius: Trial of Volar Plate Versus Dorsal Nail Plate Fixation
Acronym: RADIUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Asker og Baerum (Other)
Responsible Party: Principal Investigator, Wender Figved, Md PhD, Sykehuset Asker og Baerum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RADIUS-DVR-DNP
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Distal Radius Fractures
Keywords: Fracture; Radius; Surgery; Osteosynthesis
MeSH Terms: conditions — Wrist Fractures; Fractures, Bone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DVR (Active Comparator): Volar plate
  Interventions: Procedure: Volar plate
- DNP (Active Comparator): Dorsal nail plate
  Interventions: Procedure: Dorsal nail plate

INTERVENTIONS:
Procedure: Volar plate — Treatment with a volar plate (DVR) inserted through a volar incision of 8-10 cm over the distal radius (Henry's approach).
  Other Names: Hand Innovation, DePuy
  Arms: DVR
Procedure: Dorsal nail plate — Treatment with a dorsal nail plate (DNP) inserted through a 3-4 cm dorsal incision.
  Other Names: Hand Innovation, DePuy
  Arms: DNP

SUMMARY:
Fractures of the distal radius are one of the most common orthopaedic injuries and are associated with a high complication rate. There is a lack of clinical trials comparing the different treatment modalities of fractures of the distal radius. The purpose of this randomized trial is to assess differences in functional outcome, radiological results, and complication rate in patients 55 years and older with an unstable displaced fracture of the distal radius without articular involvement treated with a dorsal nail plate or a volar plate.

DETAILED DESCRIPTION:
Surgical treatment is needed for distal radius fractures that can not be treated with a simple plaster cast, and is indicated in a substantial amount of these patients. There is a well known correlation between a good anatomical result and a good functional outcome for the patient. The most common methods for operative fixation are external fixation with a metal frame, percutaneous pin fixation, and open surgery with insertion of a metal plate and screws on the dorsal or the volar side of the fracture. Biomechanical studies have shown differences in mechanical stability between different plate fixation systems.

The investigators are conducting this randomized trial to investigate the differences in outcome after treatment with a DVR volar plate and a DNP dorsal nail plate. The DVR volar plate follows the same principles of fixation as other volar plates using locking screws and/or pegs. It has smooth or threaded pegs that are multidirectionally placed in the distal part of the plate. The dorsal nail plate (DNP) is a relatively new implant that is inserted through a less invasive technique, with a minimum of soft tissue exposure. It is inserted through a 3-4 cm long incision on the dorsal side of the wrist and is introduced into the medullary canal. It is fixed with screws on the proximal (nail) side of the fracture and threaded or smooth locked multidirectional pegs on the distal (plate) side of the fracture. It has been suggested as a good alternative to regular plate fixation where less invasive surgery is desired. Clinical patient series have been published showing good clinical results.

There are no clinical trials comparing these two types of treatment. Therefore the investigators want to conduct a randomised controlled trial, with the purpose of finding potential differences in functional outcome for the patients.

ELIGIBILITY:
Inclusion Criteria:

* Unstable dorsally displaced fracture of the distal radius without articular involvement
* Age 55 years or older

Exclusion Criteria:

* Previous fracture of the same wrist
* More than one acute fracture (except the ulnar styloid process)
* Open fracture
* Mental impairment or unable to understand and sign an informed consent
* Fracture older than 14 days

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
DASH score | 52 weeks

SECONDARY OUTCOMES:
PRWE score | 52 weeks
EQ-5D score | 52 weeks
Grip strength | 52 weeks
Radiological result | 52 weeks
Pain VAS score (1-10) | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn Hjall, M.D., Study Chair — Asker and Baerum hospital, Norway
Locations (1):
- Asker and Baerum Hospital, Baerum, Rud, Norway